CLINICAL TRIAL: NCT05713188
Title: Clinical Investigation of the Safety of the MediSieve Magnetic Haemofiltration System in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediSieve Limited (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MediSieve FMS study
Record Dates: First submitted 2023-01-10; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Haemofiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All volunteers will receive the same treatment
  Interventions: Device: MediSieve Magnetic Haemofiltration System

INTERVENTIONS:
Device: MediSieve Magnetic Haemofiltration System — The MediSieve Magnetic Haemofiltration System is a medical device intended for use in extracorporeal clinical procedures to remove magnetic targets (e.g. malaria infected red blood cells) from a patient's bloodstream. Healthy volunteers will undergo filtration for 5 hours.

SUMMARY:
This is a single-centre, non-randomised, prospective study to assess the safety of the MediSieve blood filtration system in healthy volunteers

DETAILED DESCRIPTION:
The MediSieve Magnetic Haemofiltration System (MMHS) is a system to filter selected moieties from blood in an extracorporeal circuit by magnetic means. Initially, it is developed for the treatment of severe malaria to capture malaria-infected erythrocytes (who are weakly magnetic) to reduce the parasitaemia. However, the use of MMHS can be extended, with the use of antibodies coupled to magnetic beads, to other diseases, such as sepsis.

The MMHS has to be used first in healthy volunteers to determine its clinical safety.

To this end, 6 healthy male and female volunteers (ratio 1:1) will undergo blood filtration using the MediSieve Magnetic Haemofiltration System (without magnetic beads) for five consecutive hours. Vital signs will be continuously monitored and blood samples will be obtained serially to determine laboratory safety and immunological parameters. Furthermore, volunteers will have two follow up visits at 24 hours and 7 days post filtration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 and ≤50 years of age
* Able to comprehend and sign the Information letter and Informed Consent (IC) prior to enrolment in the study.

Exclusion Criteria:

* BMI <18.5 or >30 kg/m2
* Chronic medication use (except contraception)
* Pregnant or lactating females
* Known anaphylaxis or hypersensitivity to any (non-)investigational products or their excipients
* History or signs of severe atopic syndrome (asthma, rhinitis with medication and/or eczema)
* History or signs of haematological disease
* History or signs of thromboembolic disorders
* History of (intracranial) aneurysmal or haemorrhagic diseases
* History of any disease associated with immune deficiency
* History of cancer in the last 5 years (excluding localised skin cancer or CIS)
* History of heparin-induced thrombocytopenia (HIT)
* History of peptic / gastric ulcer disease
* Family history of haemorrhagic or thromboembolic disorders (<50 years of age)
* Thrombocytopenia (<150*109/ml) or anaemia (males: haemoglobin < 8.0 mmol/L, females: haemoglobin < 7.4 mmol/L)
* History, signs or symptoms of cardiovascular disease, in particular:

  * Prone to vagal collapse
  * History of atrial or ventricular arrhythmia
  * Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrio-ventricular block or a complete left bundle branch block
  * Hypertension (defined as RR systolic > 160 or RR diastolic > 90 mmHg)
  * Hypotension (defined as RR systolic < 100 or RR diastolic < 50 mmHg)
* Renal impairment (defined as plasma creatinine >120 μmol/L)
* Liver enzyme abnormalities (above 2x the upper limit of normal)
* Signs of infection (CRP > 20 mg/L, White Blood Count > 12x109/L or < 4x109/L)
* Clinically significant acute illness, including infections or trauma, within 1 month of the experiment day
* Participation in an experimental intervention or drug trial or donation of blood within 3 months prior to the experiment day
* Recent hospital admission or surgery with general anaesthesia within 3 months prior to experiment day
* Use of recreational drugs within 2 weeks of the experiment day
* Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse events) | Continuously starting from 2 hours prior of the start of haemofiltration until 7 days post-filtration
  Incidence of (serious) adverse events and device deficiencies during haemofiltration until 7 days post-filtration

SECONDARY OUTCOMES:
Safety (Blood pressure) | From 2 hours prior until 7 hours after start of haemofiltration.
  Systolic, diastolic and mean arterial pressure will be measured continuously using a radial artery catheter.
Safety (Heart rate) | Continuously from 2 hours prior until 7 hours after start of haemofiltration.
  Heart rate will be recorded continuously using a 3-lead ECG.
Safety (Temperature) | Every 30 minutes from 2 hours prior until 7 hours after start of haemofiltration.
  Body temperature will be assessed by using tympanic temperature measurements.
Safety (Symptoms) | Every 30 minutes from 2 hours prior until 7 hours after start of haemofiltration.
  Clinical symptoms will be scored on a Likert scale (ranging from 0 to 5) in a composite endpoint consisting of headache, nausea, shivering, muscle soreness and lower back pain. Higher numbers indicate more severe symptoms.
Safety (Immunology) | Samples will be obtained from 1 hour prior until 7 days after start of haemofiltration.
  The following plasma cytokines will be measured (pg/mL): Tumour necrosis factor (TNF), Interleukin (IL)-6, IL-8, IL-10, IL-1 receptor antagonist (IL-1RA), Monocyte Chemoattractant Protein (MCP)-1, Macrophage Inflammatory Protein (MIP)-1α, MIP-1β, Interferon-γ induced Protein (IP)-10, and Granulocyte Colony-Stimulating Factor (G-CSF)
Safety (Metal analysis) | Samples will be obtained from start of haemofiltration, and after 1 hour, 5 hours, 24 hours and 7 days.
  Plasma concentration levels of chromium and manganese will be measured in nmol/L.
Safety (Cell counts) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  Leukocytes (including differentation), erythrocytes and thrombocytes will be measured in *10^9/L.
Safety (Haemoglobin and elektrolytes) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  Haemoglobin, sodium, potassium, calcium, phosphate, magnesium, and urea will be measured in mmol/L
Safety (Haematocrit) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  Haematocrit will be measured in L/L.
Safety (Coagulation) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  Prothrombin time (PT), activated clotting time (ACT) and activated partial thromboplastin time (APTT) will be measured in seconds.
Safety (INR) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  International Normalized Ratio (INR) will be measured to assess coagulation.
Safety (Fibrinogen + albumin) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  Fibrinogen and albumin will be measured in grams/L.
Safety (Kidney function) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  Kidney function will be measured in mL/min/1.73m^2.
Safety (Markers associated with cellular damage) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  Cellular damage will be assessed by measuring Alanine Aminotransferase (ALAT), Aspartate Aminotransferase (ASAT), Lactate Dehydrogenase (LDH), Creatine kinase (CK), Alkaline phosphatase (AP)
Safety (C-reactive protein) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  C-reactive protein (CRP) will be measured in mg/L.
Safety (Creatinine and iron status) | Samples will be obtained from 2 hours prior until 7 days after start of haemofiltration.
  Creatinine, iron and total iron binding capacity (TIBC) will be measured in umol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Matthijs Kox, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided